CLINICAL TRIAL: NCT00251875
Title: Shared Online Health Records for Patient Safety and Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HS013326 (AHRQ)
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2005-11-11 (Estimated); Status verified 2005-11

CONDITIONS: Diabetes
Keywords: patient portals; electronic health records; family history; health maintenance; medications; diabetes
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Device: online health information journal

SUMMARY:
The study uses a randomized, prospective cohort design to assess the impact of shared online health records on 1) patient safety, 2) health goal adherence and outcomes, 3) documentation of family history, and 4) barriers to the adoption of patient-physician communication technology.

Hypothesis: the respective interventions will result in 1) improved patient safety 2) greater adherence to health care maintenance and chronic disease guidelines 3) more accurate documentation of family history 4) the identification of technology adoption enablers and barriers.

DETAILED DESCRIPTION:
During the first phase of the study, primary care practice patients continue to receive "usual care" while their physician's offices are using Patient Gateway, an Internet portal offering secure messaging, common requests, chart information, and health information that has already been developed. Also in this first phase, all patients using Patient Gateway will receive an electronic letter explaining the research study and a link to an electronic consent form. In addition to recruitment of subjects, phase 1 allows for baseline data to be collected.

In the second phase, study clinics will be randomized into one of two intervention "arms". Study subjects whose clinics are randomized into Arm 1 will be invited to review and comment on their medication, allergy, and diabetes information through Patient Gateway; they can then submit this information to their primary care physician for review. Those randomized into Arm 2 will report on their health maintenance status and family history and submit this information to their primary care physician through Patient Gateway prior to a scheduled visit. Chart reviews performed at the end of Phase 1 and Phase 2 will be conducted to identify differences in process measures and outcome measures between intervention and control groups.

In addition, a medication phone survey sub-study will be conducted to evaluate the effect of the new Patient Gateway features on medication management.

ELIGIBILITY:
Inclusion Criteria:

* All patients, who are enrolled in Patient Gateway, of physicians and practices participating in the study.

Exclusion Criteria:

* Any patients who are not enrolled in Patient Gateway or do not belong to a participating practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5400
Dates: Start 2005-07; Study Completion 2007-09

PRIMARY OUTCOMES:
1. ADEs
2. duration of ameliorable medication side effects
3. health goal adherence rates
4. diabetes outcomes
5. familial risk factor documentation rates
6. user satisfaction surveys
7. user metrics

CONTACTS AND LOCATIONS:
Overall Officials: Blackford Middleton, MD, MPH, MSc, Principal Investigator — Brigham & Women's Hospital, Partners HealthCare System, Inc.
Locations (10):
- United States (10):
  - Beacon Hill/Downtown Primary Care, Boston, Massachusetts
  - Bulfinch Medical Group, Boston, Massachusetts
  - Massachusetts General Hospital Women's Health Associates, Boston, Massachusetts
  - Charlestown Health Center, Charlestown, Massachusetts
  - Brigham & Women's Hospital Women's Health Center, Chestnut Hill, Massachusetts
  - Brigham & Women's Physicians Group, Chestnut Hill, Massachusetts
  - Brigham Primary Physicians at Faulkner, Jamaica Plain, Massachusetts
  - Southern Jamaica Plain Health Center, Jamaica Plain, Massachusetts
  - Brigham & Women's Hospital at Norwood, Norwood, Massachusetts
  - Revere Health Center, Revere, Massachusetts

REFERENCES:
- [Derived] Schnipper JL, Gandhi TK, Wald JS, Grant RW, Poon EG, Volk LA, Businger A, Williams DH, Siteman E, Buckel L, Middleton B. Effects of an online personal health record on medication accuracy and safety: a cluster-randomized trial. J Am Med Inform Assoc. 2012 Sep-Oct;19(5):728-34. doi: 10.1136/amiajnl-2011-000723. Epub 2012 May 3. PMID 22556186
- [Derived] Wright A, Poon EG, Wald J, Schnipper JL, Grant R, Gandhi TK, Volk LA, Bloom A, Williams DH, Gardner K, Epstein M, Nelson L, Businger A, Li Q, Bates DW, Middleton B. Effectiveness of health maintenance reminders provided directly to patients. AMIA Annu Symp Proc. 2008 Nov 6:1183. PMID 18999087
- [Derived] Grant RW, Wald JS, Schnipper JL, Gandhi TK, Poon EG, Orav EJ, Williams DH, Volk LA, Middleton B. Practice-linked online personal health records for type 2 diabetes mellitus: a randomized controlled trial. Arch Intern Med. 2008 Sep 8;168(16):1776-82. doi: 10.1001/archinte.168.16.1776. PMID 18779465